CLINICAL TRIAL: NCT01025206
Title: A Phase I Dose-Escalation Study to Determine the Safety, Pharmacokinetics, and Pharmacodynamics of BI 505, a Human Anti-Intercellular Adhesion Molecule 1 Monoclonal Antibody, in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of a Human Anti-Intercellular Adhesion Molecule-1 Monoclonal Antibody, in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BI-505-01
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2012-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; monoclonal antibody; safety; pharmacokinetic
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BI-505 (Experimental)
  Interventions: Biological: BI-505

INTERVENTIONS:
Biological: BI-505 — Anti-ICAM-1 monoclonal antibody given as a i.v infusion every second week for four weeks,

SUMMARY:
This is a first in human study which will assess the safety and tolerability of a monoclonal antibody against ICAM-1 in patients with Multiple Myeloma. The tumour response rate will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Myeloma with measurable disease after at least 2 previous regimens.
* Life expectancy > 3 months.
* Performance status ECOG < 2.

Exclusion Criteria:

* Prior antineoplastic therapy within 4 weeks prior to inclusion.
* No high dose steroids within 7 days prior to screening.
* Severe other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety assessed as Adverse Events, ECG, vital signs and clinical laboratory tests | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guido Tricot, MD, PhD, Prof., Principal Investigator — University of Utah
Locations (7):
- United States (2):
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - University of Utah Health Sciences Center, Department of Medicine, Division of Hematology, Utah Blood and Marrow Transplant and Myeloma Program, Salt Lake City, Utah
- Belgium (2):
  - AZ Sint-Jan, Bruges
  - Ghent University Hospital, Ghent
- Rigshospitalet, Copenhagen, Denmark
- Sweden (2):
  - Karolinska University Hospital, Huddinge
  - Hematology Clinic Cancer Division, Skåne University Hospital, Lund

REFERENCES:
- [Derived] Hansson M, Gimsing P, Badros A, Niskanen TM, Nahi H, Offner F, Salomo M, Sonesson E, Mau-Sorensen M, Stenberg Y, Sundberg A, Teige I, Van Droogenbroeck J, Wichert S, Zangari M, Frendeus B, Korsgren M, Poelman M, Tricot G. A Phase I Dose-Escalation Study of Antibody BI-505 in Relapsed/Refractory Multiple Myeloma. Clin Cancer Res. 2015 Jun 15;21(12):2730-6. doi: 10.1158/1078-0432.CCR-14-3090. Epub 2015 Feb 24. PMID 25712687